CLINICAL TRIAL: NCT03927976
Title: Testing the Feasibility of a Culturally-Specific Video Text Cessation Intervention With African American Quitline Callers
Brief Title: Feasibility of a Culturally-Specific Video Text Cessation Intervention With AA Quitline Callers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1Y19
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Path2Quit (Experimental): After assessment eligibility, given consent, information about text messaging will be collected and participants enrolled in the Path2Quit culturally specific text message program and feedback will be collected on their experience.
  Interventions: Behavioral: Path2Quit - culturally specific text message intervention

INTERVENTIONS:
Behavioral: Path2Quit - culturally specific text message intervention — SMS text delivers over 6 weeks with links to 20-120 second video clips from PTF. The message library contains 155 videos and assessment questions. First message is tailored to wake-up times, and the topic of the video (e.g., Never Quit Quitting) accompanies the text. Messages are pushed to participants 1-2 times/day, with 24/7 access to messages pulled from 3 keywords (HELP1, JONES, SLIP). Participants also receive inquiry texts, designed to push videos of interest/relevance to the individual. The cultural adaptations are infused throughout the video segments. Topics include deep structure: race and smoking in general, African American smoking statistics; norms for smoking; concerns about nicotine replacement/medication; family/collectivism; unique stressors; racism/discrimination, depression; co-morbid addiction; neighborhood/environmental influences; menthol cigarettes; race-specific weight issues and concerns; and working as a community against the tobacco industry.

SUMMARY:
Assess the feasibility and acceptability of delivering an mHealth tobacco intervention among state quitline enrollees.

DETAILED DESCRIPTION:
The main objective of this study is to assess the feasibility of delivering an mHealth tobacco intervention among state quitline enrollees. This will be measured through the assessment of interest and willingness to use the video text program, and the ability to receive video text messages (i.e., has technology capable of receiving and viewing video texts. At the end of the intervention, the team will assess satisfaction and perceived helpfulness of the video-text messaging program as an indication of acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American
* Enrolled in state quitlines within the past 3 months
* Have access to SMS texting

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by interest in using Path2Quit video text program | Through study completion, an average of 6-weeks.
  The program will be evaluated as feasible if 50% of those screened are eligible and interested in the video text program AND if 90% of those who are eligible and interested in the video text program will be able to engage in the program (some may need technical assistance).

SECONDARY OUTCOMES:
Acceptability of intervention in terms of its Satisfaction and perceived helpfulness: 6-Week Follow-Up Questionnaire | 6 weeks from end of intervention
  Acceptability of intervention measured through a 6-Week Follow-Up Questionnaire assessing satisfaction with Path2Quit and perceived usefulness
  Program will be evaluated as 'acceptable' if 80% of those who engage in the video text program and who answer the follow-up survey will rate their satisfaction with program and usefulness of the program at 3 or higher (on 0-7 scale where 3 indicates somewhat satisfied and somewhat useful) AND 80% rate the likelihood that they would recommend to a friend at a 3 or higher (on 0-7 point scale where 3 indicates "yes, I think so").

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States